CLINICAL TRIAL: NCT03268837
Title: Programmed Intermittent Bolus for Infusion of Local Anesthetic During Continuous Interscalene Nerve Blockade for Total Shoulder Arthroplasty: a Randomized Controlled Trial
Brief Title: Programmed Intermittent Bolus During Continuous Interscalene Nerve Block for Shoulder Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Shalini Dhir, Associate Professor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 109624
Record Dates: First submitted 2017-08-28; First posted 2017-08-31 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: Shoulder Arthroplasty; Shoulder Osteoarthritis; Pain Management
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Programmed Intermittent Bolus (PIB) (Experimental): For the experimental group, patients will receive 5 mL of the study solution as a bolus every hour via a PIB-capable infusion pump.
  Interventions: Device: Programmed Intermittent Bolus
- Continuous Infusion (Active Comparator): The control (standard care) group will receive the study solution at a rate of 5mL/h continuously via the current infusion pump.
  Interventions: Device: Continuous Infusion

INTERVENTIONS:
Device: Programmed Intermittent Bolus — The Smith CADD(R)-Solis Ambulatory Infusion Pump will be used to provide programmed intermittent bolus for the interscalene block.
  Arms: Programmed Intermittent Bolus (PIB)
Device: Continuous Infusion — The Smith CADD(R)-Solis Ambulatory Infusion Pump will be used to provide continuous infusion for the interscalene block.
  Arms: Continuous Infusion

SUMMARY:
A new infusion strategy named the 'programmed intermittent bolus' (PIB) technique delivers the hourly dose within minutes compared to the traditional infusion that delivers such dose over an hour. The PIB technique has demonstrated superior patient satisfaction and reduced local anesthetic consumption when utilized for pain control during labour and delivery. However, it is not known if the PIB technique gives any benefits during a continuous nerve block in other settings. The aim of this randomized controlled trial (RCT) is to elucidate if PIB is better than (traditional) continuous infusion for postoperative analgesia in patients receiving a continuous nerve block for total shoulder arthroplasty with respect to pain control.

DETAILED DESCRIPTION:
Local anesthetics are often given in a continuous fashion to block specific nerves after an operation for pain control. A new infusion strategy named the 'programmed intermittent bolus' (PIB) technique delivers the hourly dose within minutes compared to the traditional infusion that delivers such dose over an hour. The PIB technique has demonstrated superior patient satisfaction and reduced local anesthetic consumption when utilized for pain control during labour and delivery. However, it is not known if the PIB technique gives any benefits during a continuous nerve block in other settings. The aim of this randomized controlled trial (RCT) is to elucidate if PIB is better than (traditional) continuous infusion for postoperative analgesia in patients receiving a continuous nerve block for total shoulder arthroplasty with respect to pain control.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* American Society of Anesthesiologists (ASA) Physical Status I to III

Exclusion Criteria:

* Body mass index (BMI) > 40
* Not able to communicate in ENglish
* Unable to obtain consent
* Infection over site of placement
* Severe respiratory disease
* Cognitive or psychiatric history that would make it difficult to assess pain score
* Complex regional pain syndrome
* Chronic pain condition such as fibromyalgia, neuropathic pain
* Preoperative opioid use greater than the equivalent of morphine 50 mg PO daily
* Allergy to any of the study drug
* Coagulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Pain score on 11 point (0 - 10) numeric rating scale | FIrst 24 hour since the operation
  Postoperative pain score

SECONDARY OUTCOMES:
Local anesthetic consumption | 36 hours (or until block discontinuation)
  The total dose of local anesthetic used until the block is discontinued
Opioid consumption | 48 hours (or until discharge)
  The total amount of opioids consumed will be recorded until the patient is discharged
Side effect | through to patient discharge, on average 48 hours
  nausea, voting, pruritus
patient satisfaction | through to patient discharge, on average 48 hours
  100 mm visual analogue scale
Block complication | through to patient discharge, on average 48 hours
  persistent motor or sensory block, dyspnea, hoarseness, Horner syndrome

CONTACTS AND LOCATIONS:
Locations (1):
- St. Joseph's Health Care London, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chong MA, Wang Y, Dhir S, Lin C. Programmed intermittent peripheral nerve local anesthetic bolus compared with continuous infusions for postoperative analgesia: A systematic review and meta-analysis. J Clin Anesth. 2017 Nov;42:69-76. doi: 10.1016/j.jclinane.2017.08.018. Epub 2017 Aug 19. PMID 28830037